CLINICAL TRIAL: NCT00002507
Title: RADIATION WITH MITOMYCIN C OR PORFIROMYCIN IN THE TREATMENT OF CANCER OF THE HEAD AND NECK AREA
Brief Title: Radiation Therapy and Chemotherapy in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000078021; YALE-HIC-6611; NCI-V92-0190
Record Dates: First submitted 1999-11-01; First posted 2004-08-10 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2000-06

CONDITIONS: Carcinoma of Unknown Primary; Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage I squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; newly diagnosed carcinoma of unknown primary; recurrent carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Mitomycin; Porfiromycin; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: mitomycin C
Drug: porfiromycin
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether combining mitomycin or porfiromycin with radiation therapy is more effective in treating patients with head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus either mitomycin or porfiromycin in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of mitomycin vs. porfiromycin as an adjunct to radiotherapy for the treatment of epidermoid carcinomas of the head and neck.

OUTLINE: Randomized study. Arm I: Radiotherapy plus Single-Agent Chemotherapy. Irradiation of involved head and neck sites by external-beam radiotherapy (EBRT) alone (source not specified), brachytherapy alone (using permanent or removable radiation sources), or both; plus Mitomycin, MITO, NSC-26980. Arm II: Radiotherapy plus Single-Agent Chemotherapy. Radiotherapy as in Arm I; plus Porfiromycin, NSC-56410.

PROJECTED ACCRUAL: Approximately 200 patients will be entered over 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven epidermoid carcinoma of the following head and neck sites: Hypopharynx Oral cavity Larynx Oropharynx Nasopharynx Unknown primary origin with positive head and neck nodes TNM Stages I-IV or recurrent disease with no distant metastases, i.e.: T1 N0 M0 T1 N1-3 M0 T2-4 any N M0 T0 N1-3 M0 No carcinoma of the true vocal cord or other condition with greater than 90% probability of cure

PATIENT CHARACTERISTICS: Age: 20 to 80 Performance status: Not specified Hematopoietic: WBC at least 3,000 Platelets at least 100,000 Hct at least 25% Hepatic: Bilirubin less than 1.5 mg/dl Renal: Creatinine less than 2 mg/dl OR BUN less than 40 mg/dl Other: No other serious, life-threatening illness No second malignancy within 5 years except nonmelanomatous skin cancer outside the planned radiotherapy field

PRIOR CONCURRENT THERAPY: At least 3 years since chemotherapy No prior radiotherapy to areas of current disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-11; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J. Fischer, MD, PhD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States